CLINICAL TRIAL: NCT04141540
Title: Translational 22q11.2:"Molecular Variants Associated With Schizophrenia: Differential Analysis of Monozygotic Twins With Variable Phenotypic 22q11.2 Microdeletional Syndrom"
Brief Title: Molecular Variants Associated With Schizophrenia: Differential Analysis of Monozygotic Twins With Variable Phenotypic 22q11
Acronym: CSRK05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A00852-55
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-06

CONDITIONS: Di George Syndrome
Keywords: 22q11.2 Microdeletional
MeSH Terms: conditions — DiGeorge Syndrome | interventions — Molecular Docking Simulation

STUDY DESIGN:
Intervention Model Description: It's a study with a comparative monocentric cross-sectional analysis model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groupe "Twin 1" (Other): Twin 1 with psychotic symptoms (PANSS +) Molecular analyses 1
  Interventions: Genetic: Molecular analyses
- Groupe "Twin 2" (Other): Twin 2 without psychotic symptoms (PANSS +) Molecular analyses 2
  Interventions: Genetic: Molecular analyses

INTERVENTIONS:
Genetic: Molecular analyses — Comparaison of the molecular profil between two monozygotic twins carrying a deletion 22q11.2

SUMMARY:
The 22q11.2 microdeletion syndrome (22q11.2DS) is a rare disease with a psychiatric phenotype. Indeed, the diagnosis of schizophrenia is made in 5 to 10% of adolescents and 25 to 40% of adults carrying the 22q11DS. Thus, although this pathology has been able to provide a genetically homogeneous model for the study psychosis etiology, it is not currently possible to establish a link between genomic rearrangement and psychotic symptoms. However, this robust model of genetic vulnerability could provide us a lot of translational informations about schizophrenia genetics. To go furthermore, twin studies have provided us precious data for the study of hereditary diseases. Combining this two approaches, the translational 22q11.2 project proposes a molecular study of two monozygotic 22q11.2DS twins discordant for the psychiatric phenotype -one carrying schizophrenia and the other having no psychiatric symptoms-.

DETAILED DESCRIPTION:
The main objective of the study is to propose a whole exome sequencing (WES), pan-genomic in whole genome sequencing (WGS), transcriptomic, epigenomic and intestinal microbiome approaches in order to determine specific molecular basis of psychotic symptoms in 22q11.2DS.

ELIGIBILITY:
Inclusion Criteria:

* • Sisterhood of monozygotic twins diagnosed with de novo 22q11.2DS is confirmed by CGH array and discordant for the psychiatric phenotype

Exclusion Criteria:

* • Refusal to use data for research purposes

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Whole exome sequencing | 6 months
  Searching for mosaic genetic variations that may have occurred secondarily to conception

SECONDARY OUTCOMES:
Transcriptome | 6 months
  two methods of mRNA extraction will be used: from the establishment of lymphoblastoid lines and from whole blood collected on paxgene® tube. After depletion of ribosomal RNA, the RNAs will be converted into complementary DNAs and libraries will be made using 100 to 200ng of total RNA. Libraries will be sequenced in a paired-end to generate 80 million reads per sample. The data will be analyzed with the HTSeq suite to count the number of reads associated with each gene annotated in the latest version of the genome. The DESeq bioconductor suite will be used to normalize the expression. A study to identify differentially expressed genes will be performed with this tool and GFold. Genes showing statistically significant differential expression will be validated by RT-qPCR
Methylome | 6 months
  This analysis will be carried out in collaboration with " L'hôpital de Sainte Anne2 (Inserm UMR_S894 "Physiology of psychiatric diseases" - Professor Marie-Odile KREBS). The DNA will be extracted from whole blood collected on paxgene® tube. The methylation of the entire genome of twin siblings will be studied by the Infinium MethylationEPIC BeadChip chip (Illumina) that covers 850,000 CpG and the set of genes after bisulfite DNA processing. The statistical analysis of the methylation differences will be carried out with the R software (minfi and ChAMP packages) in order to highlight the DMP (Differentially Methylated Probes) as well as the DMR (Differentially Methylated Regions, probes contigues).
Microbiotic DNA | 6 months
  A quantitative metagenomic analysis will be carried out on the basis of a sequencing of the genetic material extracted from the intestinal microbiome in the stools of the two twins
Positive And Negative Syndrome Scale (PANSS) | 6 months
  Scale of evaluation of positive and negative syndromes of schizophrenic symptomatology.The patient is rated from 1 to 7 on 30 different symptoms based on the interview as well as reports of family members or primary care hospital workers.As 1 rather than 0 is given as the lowest score for each item, a patient can not score lower than 30 for the total PANSS score. Scores are often given separately for the positive items, negative items, and general psychopathology.
Mini-International Neuropsychiatric Interview (MINI) | 6 months
  The modalities for answering all the Mini-International Neuropsychiatric Interview (MINI)questions are "YES" or "NO". If the answers to these filter questions are positive, the following ones are asked allowing to validate or invalidate the diagnosis concerned.
Hospital Anxiety and Depression Scale (HADS) | 6 months
  The Hospital Anxiety and Depression Scale (HADS) is an instrument for detecting anxiety and depressive disorders. It has 14 listed items from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), allowing thus obtaining two scores (maximum score of each score = 21).

CONTACTS AND LOCATIONS:
Overall Officials: DEMILY CAROLINE, MD PH.D, Principal Investigator — Centre Hospitalier le Vinatier & CNRS UMR 5229 (BRON, France)
Locations (1):
- Hopital Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No